CLINICAL TRIAL: NCT01156779
Title: A Dose Block-randomized, Double-blind, Placebo-controlled, Dose-escalating, Phase I Study to Evaluate Safety and Pharmacokinetics/Pharmacodynamics of DA-3091 After Subcutaneous Injection in Healthy Male Subjects
Brief Title: Study to Evaluate Safety and PK/PD of DA-3091 in Healthy Male Subjects
Acronym: SR-Exenatide
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dong-A Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Dong-A ST Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DA3091_DM_I
Record Dates: First submitted 2010-07-02; First posted 2010-07-05 (Estimated); Last update posted 2013-08-13 (Estimated); Status verified 2013-08

CONDITIONS: Diabetes Mellitus
Keywords: SR-Exenatide
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DA-3091 (Experimental): SR-exenatide
  Interventions: Drug: SR-exenatide
- Placebo of DA-3091 (Placebo Comparator): Placebo
  Interventions: Drug: SR-exenatide

INTERVENTIONS:
Drug: SR-exenatide — Emulsion 0.5mg,1mg,2mg,4mg dosage (Dose-escalation) Single injection
  Other Names: DA-3091

SUMMARY:
This Phase I clinical study is to evaluate the safety and tolerance of DA-3091 and to characterize the pharmacokinetic/pharmacodynamic of DA-3091 in healthy male subjects

DETAILED DESCRIPTION:
This is a phase I dose escalation study. To meet the clinical objectives, we are using a two-part approach. In part I, 4 subjects are injected 0.5mg dose of DA-3091 or placebo(Single/Subcutaneous Injection). After completion of part I study, we are reporting data about safety to IDMC. In part II, 8 subjects per group are injected 1mg, 2mg, 4mg of DA-3091 or placebo through dose escalating protocol. The ratio of DA-3091 and placebo is 3:1.

ELIGIBILITY:
Inclusion Criteria:

1. Age : 20 ~ 45 years old
2. Healthy Male
3. Body weight : ≥50kg and Ideal body weight ± 20%
4. Informed consent

Exclusion Criteria:

1. Clinically significant medical history
2. Acute or Chronic pancreatitis
3. Clinically significant hypersensitivity of Drugs
4. Clinically significant cutaneous disorder
5. History of administration of exenatide
6. Disorder of blood pressure
7. History of drug abuse

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2010-07; Primary Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Assessment of safety | 84 days
  1. Adverse Events
  2. Laboratory Results
  3. Vital sign, Physical Examination, EKG

SECONDARY OUTCOMES:
Pharmacokinetics and Pharmacodynamics | PK : 84 days / PD : 42days
  PK : Cmax, Tmax, AUClast PD : Glucose, Insulin, Glucagon, C-peptide in blood sample

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Sang Yu, M.D., Ph.d, Principal Investigator — Seoul National University Hospital
Locations (1):
- Clinical Trial center, Clinical Research institute, Seoul National University Hospital, Seoul, South Korea